CLINICAL TRIAL: NCT03853811
Title: Customized Orthosis for Children With Clubfoot Following Ponseti Casting
Brief Title: Customized Orthosis for Children With Clubfoot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Scott Van Valin, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1246407
Record Dates: First submitted 2019-01-20; First posted 2019-02-26 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Congenital Talipes Equinovarus
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitchell Shoe + AFO (Experimental): Group will receive standard Mitchell shoes along with the custom orthotic insert.
  Interventions: Device: Ankle Foot Orthosis (AFO)
- Standard Mitchell Shoe (Control - Standard Treatment) (No Intervention): Group will receive standard treatment which includes bracing with standard Mitchell shoes (no custom orthotic). Patients would receive this treatment regardless of study participation.

INTERVENTIONS:
Device: Ankle Foot Orthosis (AFO) — The intervention group will receive the custom AFO to use in their standard Mitchell shoe.
  Arms: Mitchell Shoe + AFO

SUMMARY:
This study will examine the use of a novel customized Ankle Foot Orthosis (AFO), created using 3D scanning, with children being treated for clubfoot. The AFO is inserted in the standard Mitchell shoe during bracing, following Ponseti casting. The investigators hypothesize that following Ponseti casting, the implementation of customized AFOs with Ponseti bracing will improve patient compliance and functional outcomes as well as lead to fewer relapses in comparison to the standard bracing with Mitchell shoes.

ELIGIBILITY:
Inclusion Criteria:

* less than 12 months old (no age minimum)
* no neuromuscular disease involved
* treated by Ponseti casting
* idiopathic bilateral or unilateral clubfoot
* no other congenital foot deformity
* no previous open surgeries to treat the deformity

Exclusion Criteria:

* patients with prior surgical treatment
* not treated by Ponseti casting
* an underlying syndrome
* neurological disorder

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Assessment of Functional Outcomes of Bracing Treatment Using Dimeglio Scores | Collected when visit where cast is applied, visit when cast is removed, then at 2 weeks, 12 weeks, 24 weeks of bracing
  Assessed using changes in Dimeglio Scores. The Dimeglio scoring system uses a 20-point system (20 being the most severe and <5 as benign) by assessing four parameters. The severity of the deformity is then assigned a grade of I-IV with IV being the most severe. (A score of <5 is given a grade of I, =5<10 is grade II, =10<15 is grade III, and =15<20 is grade IV)
Time Spent in Brace to Assess Brace Compliance | 24 weeks (from start of bracing treatment)
  Measured with sensor placed in Mitchell shoe
Assessing Treatment Factors that Impact Brace Compliance with Parental Questionnaires | 24 weeks (from start of bracing treatment)
  Assessing reasons for poor compliance with parental questionnaires. The questionnaires ask questions about casting, occurrences of skin lesions, history of treatments, bracing information, reasons for not using brace, and brace slippage

SECONDARY OUTCOMES:
Assessing Demographic Factors that Impact Brace Compliance with Parental Questionnaire | 24 weeks (from start of bracing treatment)
  The initial questionnaire asks questions about parental demographics to determine what factors may influence brace treatment compliance

CONTACTS AND LOCATIONS:
Overall Officials: Scott Van Valin, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT03853811/Prot_SAP_000.pdf